# Nasal high frequency oscillation ventilation versus nCPAP to reduce post-extubation pCO<sub>2</sub> in very low birth weight infants: a randomized controlled trial

# **Objectives**

To investigate whether nasal high frequency oscillation ventilation (nHFOV) immediately after extubation reduces the  $paCO_2$  in comparison with nasal continuous positive airway pressure (nCPAP) at 72 hours after extubation in very low birth weight infants (VLBWs).

### Protocol/Methods

### 1. Trial design

Randomized controlled clinical trial of nHFOV versus nCPAP immediately after extubation.

### 2. Participants

Eligibility criteria

- Gestational age <32+0 weeks
- Birth weight <1500 g
- Received mechanical ventilation via an endotracheal tube for ≥120 h
- Caffeine treatment according to unit guidelines
- Arrival at the preset extubation criteria:
  - o Time-cycled, pressure-controlled ventilation:

 $PIP \le 22 \text{ cm H}_2O$ ,  $PEEP \le 6 \text{ cm H}_2O$ ,

 $F_iO_2$  25-40% to maintain SpO<sub>2</sub> at 90-94%.

 $paCO_2 < 65 \text{ mmHg with pH} > 7.2$ 

o Volume guarantee ventilation:

Working  $P_{peak} \le 22 \text{ cm H}_2O$ ,  $PEEP \le 6 \text{ cm H}_2O$ 

F<sub>i</sub>O<sub>2</sub> 25-40% to maintain SpO<sub>2</sub> at 90-94%.

 $paCO_2 < 65 \text{ mmHg with pH} > 7.2$ 

o High frequency oscillation ventilation: set  $P_{mean} \le 12$  cm  $H_2O$ , Amplitude  $\le 30$  cm  $H_2O$ 

F<sub>i</sub>O<sub>2</sub> 25-40% to maintain SpO<sub>2</sub> at 90-94%.

 $paCO_2 < 65 \text{ mmHg with pH} > 7.2$ 

• Decision of the attending clinician to extubate

## Exclusion criteria

- Major congenital malformation requiring surgery (e.g. esophageal atresia, diaphragmatic hernia, abdominal wall defect)
- Duct-dependent congenital heart disease
- Neuromuscular disease
- Participation in another RCT
- Death before reaching the eligibility criteria
- Hydrocortisone treatment at the time of enrolment
- Chronological age >28 days

## 3. Study settings

Two universitarian tertiary neonatal intensive care units in Berlin.

### 4. Intervention

Application of nHFOV or nCPAP immediately after extubation from endotracheal HFOV or from conventional ventilation.

### • Equipment:

- Devices used for endotracheal ventilation, nHFOV and nCPAP: Leoni Plus (Heinen und Löwenstein, Germany) or VN 500 (Dräger, Germany)
- Interfaces: Endotracheal tubes (Vygon, France; Portex, Smiths Medical, UK) for endotracheal ventilation. Binasal prongs (Fisher & Paykel, New Zealand) for nHFOV and nCPAP.
- o Humidifier: MR 850 AGU (Fisher & Paykel, New Zealand)
- Primary intervention:
  - o Extubation by withdrawing the endotracheal tube without sustained inflation
  - o nHFOV group: immediately after extubation, apply nHFOV via binasal prongs. Set frequency at 10 Hz, I:E ratio 33:66, Amplitude 20 cm H<sub>2</sub>O, Pm 8 cm H<sub>2</sub>O, flow automatic (7 l/min).
    - Set F<sub>i</sub>O<sub>2</sub> to maintain SpO<sub>2</sub> at 90-94%.
  - nCPAP group: immediately after extubation, apply nCPAP via binasal prongs.
    Set CPAP level at 8 cm H<sub>2</sub>O, flow 7 l/min.
    Set F<sub>i</sub>O<sub>2</sub> to maintain SpO<sub>2</sub> at 90-94%.
- Weaning of non-invasive respiratory support:
  - o The weaning process is left to the discretion of the attending physician.
  - Once the infant is considered stable on nHFOV, intermittent or permanent weaning to nCPAP is allowed.
  - o Once the infant is considered stable on nCPAP, intermittent or permanent weaning to high flow nasal cannula is allowed.
- Increasing non-invasive respiratory support:
  - O Increasing non-invasive respiratory support is left to the discretion of the attending physician. The following settings are allowed in the nHFOV- and nCPAP-group, respectively.
  - o nHFOV group:
    - Maximum amplitude 30 cm H<sub>2</sub>O, minimum frequency 9 Hz.
    - Maximum set P<sub>mean</sub> 8 cm H<sub>2</sub>O.
  - o nCPAP group:
    - Maximum CPAP level 8 cm H<sub>2</sub>O, maximum flow 8 l/min.
- Definition of treatment failure (infant meets at least one criterion):
  - Sustained pCO<sub>2</sub> >80 mmHg and pH <7.20 confirmed by arterial or capillary blood gas analysis in spite of optimized non-invasive respiratory support with maximum settings as defined above.
  - $\circ$  F<sub>i</sub>O<sub>2</sub> >0.6 to maintain SpO<sub>2</sub> at 90-94% in spite of optimized non-invasive respiratory support with maximum settings as defined above.
- Reintubation:
  - Study patients may be intubated at any time due to clinical considerations (with or without reaching a criterion of "treatment failure", as defined above).
- "Rescue-nHFOV" for infants in the nCPAP-group who "fail" nCPAP (defined as reaching a criterion of "treatment failure", as defined above), but do not need immediate reintubation:
  - o Trial of nHFOV via binasal prongs.
  - o Choice of nHFOV settings are at the discretion of the attending clinician.
- "Rescue treatment" for infants in the nHFOV-group who "fail" nHFOV (defined as reaching a criterion of "treatment failure", as defined above), but do not need immediate reintubation:

- Choice of non-invasive respiratory support for the "rescue treatment" (e.g. nIPPV, nHFOV) and ventilator settings are at the discretion of the attending clinician.
- Planned data collection to document the respiratory support provided in the nCPAP- and the nHFOV-group:
  - o Blood gas result before extubation (pH, paO<sub>2</sub>, paCO<sub>2</sub> and BE).
  - $\circ$  Ventilator settings before extubation (mode and  $F_iO_2$  in all patients; set  $P_{mean}$  during HFO; PIP and PEEP during time-cycled, pressure-controlled ventilation; working  $P_{peak}$  and PEEP during volume guarantee ventilation).
  - O Documentation of non-invasive respiratory support, including settings of nHFOV and/or nCPAP every 24h during the first 3 days after extubation and at 7 days after extubation (mode, set mean nHFOV pressure, frequency, amplitude; CPAP level; flow, F<sub>i</sub>O<sub>2</sub>), and after switch to "rescue treatment" or "rescue-nHFOV", if applicable.

### 5. Outcomes

- Primary outcome:
  - o paCO<sub>2</sub> at 72 h (timeframe: 64 h to 80 h) after extubation
- Secondary outcomes:
  - o pH, paO<sub>2</sub>, paCO<sub>2</sub>, BE at 2 h (timeframe: within first 6 h) after extubation
  - o pH, paO<sub>2</sub>, BE at 72 h (timeframe: 64 h to 80 h) after extubation
  - Successful extubation (defined as spontaneous breathing in the assigned treatment group for ≥72h without being reintubated or reaching the criterion of "treatment failure", as defined above)
  - Treatment failure (defined as reaching the criterion of "treatment failure", as defined above, within the first 7 days after extubation)
  - o Reintubation within the first 7 days after extubation
  - Adverse effects observed after extubation: documented episodes of airway obstruction due to highly viscous secretions, IVH III°-IV° (Papile), surgical NEC, pneumothorax, pulmonary interstitial emphysema, mild BPD (Jobe), PDA requiring surgical closure, ROP requiring laser treatment and/or injection of bevacizumab, PVL
  - Respiratory support: total duration of mechanical ventilation, total duration of supplemental oxygen, number of infants discharged with home oxygen
- Additional secondary outcomes for those infants who received "rescue treatment":
  - o pH, paO<sub>2</sub>, paCO<sub>2</sub>, BE at 2 h (timeframe: within first 6 h) after switch to "rescue" therapy
  - Successful rescue (defined as spontaneous breathing for ≥72h after starting "rescue" therapy, without reaching the criterion of "treatment failure", as defined above)
- Follow-up study:
  - o Lung function testing at 52 weeks' corrected gestational age.

### 6. Sample size

Assuming a variability of the paCO<sub>2</sub> as previously reported for difficult-to-wean preterm infants in our unit (Czernik C, *J Matern Fetal Neonatal Med* 2012) and a reintubation rate of 21% within 72 h after extubation, we calculated a sample size of 28 patients in each study arm to detect a difference in the paCO<sub>2</sub> of 7 mmHg between the study groups, using a two-sided significance of 0.05 and a power of 0.8.

# 7. Interim analyses and stopping guidelines

An independent statistician performs an interim-analysis on the primary and secondary endpoints once 50% of the patients are randomized and outcome data is available.

# 8. Randomization: sequence generation

Sequence generation by an independent statistician and a study nurse.

# 9. Randomization: type

Block randomization using at least two different block sizes, stratification by center.

# 10. Randomization: allocation concealment mechanism

Sequentially numbered opaque sealed envelopes. Patients are randomized immediately before extubation.

# 11. Registration of the trial

clinicaltrials.gov

Document dated 03-13-2012 Document translated 01-15-2015